CLINICAL TRIAL: NCT05348382
Title: The Efficacy and Safety of Intradermal Acupuncture for Acute Herpes Zoster: Study Protocol for a Randomized Controlled Trial
Brief Title: The Efficacy and Safety of Intradermal Acupuncture for Acute Herpes Zoster
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Hantong Hu, Attending doctor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022ZB184
Record Dates: First submitted 2022-04-17; First posted 2022-04-27 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Herpes Zoster
Keywords: herpes zoster; intradermal acupuncture; infrared thermography; clinical trial
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intradermal acupuncture group (Experimental): Points around the herpes zoster sites (about 1 cm peripherally) are selected for intradermal acupuncture (IDA) encircled needling. Meanwhile, intradermal acupuncture is also performed in Ashi acupoints in the distribution area of herpes zoster.
  Interventions: Procedure: Intradermal acupuncture
- Sham intradermal acupuncture group (Sham Comparator): Sham intradermal acupuncture will be implemented in the same acupoints as the intradermal acupuncture group using pseudo-intradermal needling.
  Interventions: Procedure: Sham intradermal acupuncture

INTERVENTIONS:
Procedure: Intradermal acupuncture — In addition to basis standard pharmacological treatments, intradermal needles will be inserted in each selected acupoint and retained in place for 48 hours. Points around the herpes zoster sites (about 1 cm peripherally) are selected for intradermal acupuncture (IDA) encircled needling. Meanwhile, intradermal acupuncture is also performed in Ashi acupoints in the distribution area of herpes zoster. The operator will tear off the adhesive tape of intradermal needles and stick them on the selected acupoints, and then apply pressure on intradermal needles over the selected acupoints perpendicularly according to the patient's tolerance. In addition, patients will be instructed to press the intradermal needles 4 times per 24 hours throughout the needle retention period, with the aim to increase stimulation for treatment enhancement, each time lasting around 30 seconds.
  Arms: Intradermal acupuncture group
Procedure: Sham intradermal acupuncture — In addition to basis standard pharmacological treatments, sham intradermal acupuncture will be implemented in the same acupoints as the intradermal acupuncture group using pseudo-intradermal needling. Additionally, participants in the sham intradermal acupuncture group will be treated in another room to avoid direct communications with subjects in the IDA group.
  Arms: Sham intradermal acupuncture group

SUMMARY:
Herpes zoster (HZ), also commonly known as shingles, is characterized by a bandlike rash in the dermatome that corresponds to the affected nerve. Pain is prevalent in HZ patients, which may be provoked by light touch. Postherpetic neuralgia (PHN) is one of the most common complications of HZ and it is generally intractable to treat.

At present, common treatment methods for HZ include anti-inflammatory, antiviral, analgesic, and neuroleptic regimens. Nevertheless, the application of these therapies can sometimes be limited by side effects. In this scenario, it is urgent to seek alternative non-pharmacological therapies for treating HZ.

Intradermal acupuncture (IDA) is a common type of acupuncture. By retaining the needles for a much longer duration than other common modalities of acupuncture, IDA can prolong the sustained effect of acupuncture. In addition, characterized by mild pain during the insertion of intradermal needles, IDA is more suitable for patients who fear conventional acupuncture and it is also easy to operate by practitioners. Therefore, concerning the treatment of pain conditions, such as acute HZ, it may have certain advantages over conventional acupuncture. Thus, The aim of this trial is to evaluate the efficacy and safety of IDA for acute HZ.

DETAILED DESCRIPTION:
This randomized controlled trial will enroll 72 eligible patients with acute herpes zoster. Participants who are confirmed eligibility will be randomly allocated to either the IDA group or the sham IDA group in a 1:1 ratio. The duration of the trial will include two study phases, including a 1-month intervention phase and a 3-month follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

1. Participants have confirmed diagnosis of herpes zoster;
2. Herpes zoster is in the acute stage and participants have not yet received antiviral treatment or analgesic treatment;
3. 18≤Age≤80 years, regardless of gender;
4. Significant pain with a visual analog scale (VAS) score ≥ 4;
5. Absence of other diseases causing skin temperature change;
6. Participants can understand the study procedure and agree to sign the informed consent form.

Exclusion Criteria:

1. Participants have some specific types of herpes zoster, such as disseminated herpes zoster; or herpes zoster is located on regions that are not suitable for intradermal acupuncture, such as the head, face, or perineum.
2. Pregnant or lactating subjects;
3. Participants have scar constitution or have severe cardiovascular, hepatic, renal, and hematopoietic system diseases that result in bleeding tendency, thereby making them unsuitable for intradermal acupuncture;
4. Participants with severe cognitive impairment who are unable to fully understand the trial protocol;
5. Participants are taking part in other trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | at baseline (pre-treatment), at 1 month after intervention, at 3-month follow-up
  The pain intensity is assessed using the 10-point Visual Analog Scale (VAS)
Stopping time of herpes zoster | through study completion (up to 4 months)
  the number of days required for herpes zoster to stop increasing
Crusting time of herpes zoster | through study completion (up to 4 months)
  the number of days required for herpes zoster crusting
Removal time of herpes zoster scabs | through study completion (up to 4 months)
  the number of days required for all herpes zoster scabs to be completely shed
Change in the temperature of regions of interest (ROIs) | at baseline (pre-treatment), at 1 month after intervention, at 3-month follow-up
  The temperature of ROIs will be assessed by infrared thermography.
Incidence rate of postherpetic neuralgia (PHN) | at 3-month follow-up
  The incidence rate of PHN will be assessed by calculating the percentage of patients who suffer from PHN

SECONDARY OUTCOMES:
Change in quality of life | at baseline (pre-treatment), at 1 month after intervention, at 3-month follow-up
  The 36-item Short Form Health Survey (SF-36) will be utilized to assess the quality of life.
Adverse events | through study completion (up to 4 months)
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Hantong Hu, MD, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (2):
- China (2):
  - the Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang
  - The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu H, Shen Y, Li X, Tian H, Li X, Li Y, Cheng Y, Wu L, Han D. Efficacy of Electroacupuncture Therapy in Patients With Postherpetic Neuralgia: Study Protocol for a Multicentre, Randomized, Controlled, Assessor-Blinded Trial. Front Med (Lausanne). 2021 May 21;8:624797. doi: 10.3389/fmed.2021.624797. eCollection 2021. PMID 34095161
- [Background] Fleckenstein J, Kramer S, Hoffrogge P, Thoma S, Lang PM, Lehmeyer L, Schober GM, Pfab F, Ring J, Weisenseel P, Schotten KJ, Mansmann U, Irnich D. Acupuncture in acute herpes zoster pain therapy (ACUZoster) - design and protocol of a randomised controlled trial. BMC Complement Altern Med. 2009 Aug 12;9:31. doi: 10.1186/1472-6882-9-31. PMID 19674449
- [Derived] Hu H, Cheng Y, Wu L, Han D, Ma R. Investigating the Therapeutic Effect of Intradermal Acupuncture for Acute Herpes Zoster and Assessing the Feasibility of Infrared Thermography for Early Prediction of Postherpetic Neuralgia: Study Protocol for a Randomized, Sham-Controlled, Clinical Trial. J Pain Res. 2023 Apr 26;16:1401-1413. doi: 10.2147/JPR.S406841. eCollection 2023. PMID 37131531